CLINICAL TRIAL: NCT06124326
Title: A Single Group Study to Evaluate the Effects of a Supplement on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rael (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20338
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Premenstrual Syndrome Supplement (Experimental): During the first menstrual cycle, participants will take the supplement as needed (pro re nata) when they feel symptoms of PMS, such as cramping or bloating.
  For the second and third menstrual cycles, Participants will take 2 capsules per day with water for 1 week, starting 4 days before their menstrual cycle and finishing on Day 3 of their cycle.
  Interventions: Dietary Supplement: Premenstrual Syndrome Supplement

INTERVENTIONS:
Dietary Supplement: Premenstrual Syndrome Supplement — Ginger, Curcumin, Organic Turmeric, Black Pepper, Magnesium, Zinc, Vitamin B6, Vitamin D.

SUMMARY:
This is a virtual single-group study that will last three menstrual cycles (approximately 12 weeks). During the first menstrual cycle, participants will take the supplement as needed (pro re nata) when they feel symptoms of PMS, such as cramping or bloating. For the second and third menstrual cycles, Participants will take 2 capsules per day with water for 1 week, starting 4 days before their menstrual cycle and finishing on Day 3 of their cycle. Questionnaires will be completed at the following time points:

* Baseline
* Day 7 of their first cycle during the trial (After using the product PRN during their period)
* 4 days before their second period during the trial (After using the product PRN for the previous month)
* Day 3 of their second period during the trial (After using the product for 7 days straight)
* Day 3 of their third period of the trial (After using the product for 7 days straight)

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-40
* Self-reported moderate discomfort during menstruation related to pelvic cramps, bloating, fatigue, or mood swings.
* Self-reported symptoms during their menstrual cycle with gas, heartburn, and acid reflux
* Generally healthy - don't live with any uncontrolled chronic disease
* Has a menstrual cycle between 21 and 35 days in length
* Able to predict their menstrual cycle and timing of their menstruation

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Current use of any blood thinning medication
* Anyone with known severe allergic reactions.
* Women who are pregnant, breastfeeding, or attempting to become pregnant
* Unwilling to follow the study protocol.
* Anyone with a diagnosis of a condition relating to the menstrual cycle or reproductive system? e.g., polycystic ovary syndrome (PCOS), premenstrual dysphoric disorder (PMDD), endometriosis, etc.
* Anyone currently on hormonal birth control, or has been on hormonal birth control in the last 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Changes in pelvic cramps. | Baseline to Week 12
  Participants will complete study-specific questionnaires. Questionnaires will include 5-point Likert scale, with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in energy levels. | Baseline to Week 12
  Participants will complete study-specific questionnaires. Questionnaires will include 5-point Likert scale, with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in overall mood. | Baseline to Week 12
  Participants will complete study-specific questionnaires. Questionnaires will include 5-point Likert scale, with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in bloating. | Baseline to Week 12
  Participants will complete study-specific questionnaires. Questionnaires will include 5-point Likert scale, with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").
Changes in gastrointestinal discomfort. | Baseline to Week 12
  Participants will complete study-specific questionnaires. Questionnaires will include 5-point Likert scale, with 5 representing the most favorable/best outcome (e.g., "Not at all") and 1 representing the least favorable/worst outcome (e.g., "Severe").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided